CLINICAL TRIAL: NCT00726206
Title: Correlation Between the Analysis of the Rapid Cortical Oscillations, the General Movements of the Preterm's and the Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2008-A00062 53; 2008-02
Record Dates: First submitted 2008-07-30; First posted 2008-07-31 (Estimated); Last update posted 2014-08-28 (Estimated); Status verified 2014-08

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other): Recording of the movements Recording of the electroencephalogram
  Interventions: Other: Electroencephalogram, recording the movements

INTERVENTIONS:
Other: Electroencephalogram, recording the movements — Electroencephalogram, recording the movements of the child, RMI, Transfontanel Imaging

SUMMARY:
The general movement and the electroencephalogram analysis of the preterm have a high predictive value of the neuro-developmental outcome of the infants.

DETAILED DESCRIPTION:
Compare the technical and the predictive characteristics of the qualitative analysis of the spontaneous motility with those of actual exams of reference diagnosis : magnetic resonance imaging, electroencephalogram and transfontanellar imaging.

ELIGIBILITY:
Inclusion Criteria:

* Children been born between 15/01/08 and 15/01/10
* children whose term is lower than 28 weeks of amenorrhoea

Exclusion Criteria:

* Born child superior to 28 weeks of amenorrhoea
* presenting child a genic syndrome, an evolutionary neurological disease, a pathology malformative

Max Age: 23 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 44 (Actual)
Dates: Start 2008-07; Primary Completion 2010-08 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
To prove the predictive value of the " Deltas Brushes " triggered by hand or foot stimulation in correlation with the general movement analysis in the cerebral palsy diagnosis. | 36 months

SECONDARY OUTCOMES:
To prove that the general movement of the preterm increases the predictive value the actual monitoring of the preterm's in the diagnosis of cerebral palsy. | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Catherine GIRE, MD, Principal Investigator — Assistance Publique des Hopitaux de Marseille
Locations (1):
- Service de Médecine Infantile et Néonatologie, CHU Nord, Marseille, France